CLINICAL TRIAL: NCT00612131
Title: Medical Residents Performance in Maximum Barrier Precautions During Central Venous Catheter Placement: Effect of Simulation-Based Training
Brief Title: Medical Residents Performance: Effect of Simulation-Based Training
Status: Completed | Type: Observational
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Other Study IDs: 07-125
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2007-09

CONDITIONS: Healthy
Keywords: medical residents PGY 2 and 3

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
I Hypothesis:

1. Simulation-based training in maximal barrier precaution technique during central venous catheter (CVC) placement is superior to general videotape-based training
2. Baseline performance in maximal barrier precaution technique of PGY 2 and 3 Medical residents, certified in CVC placement, is poor
3. PGY 2 and 3 medical residents have low self-perceived confidence in mastering maximal barrier precaution technique during central venous catheter (CVC) placement
4. PGY 2 and 3 medical residents undergoing simulation-based training in maximal barrier precaution technique during central venous catheter (CVC) placement have good recall after 3 months

DETAILED DESCRIPTION:
Central line associated bloodstream infection (CL-ABI) is an important and preventable cause of nosocomial infections and is responsible for considerable morbidity and mortality. It is estimated that 5 to 26% of patients experience an infectious complication from their central venous catheter [1]. In the United States, it is estimated that nearly 50,000 patients develop central line associated bloodstream infections in the ICUs annually, at a rate of approximately 5 infections per 1000 catheter days [2] and as many as 15,000 deaths annually. Central line associated bloodstream infections are also associated with increased hospital and ICU lengths of stay in the ICU (2). Estimates of the cost of CL-ABI to hospitals range from $25,000 to $65,000 per patient [3, 4].

The Centers for Disease Control have published guidelines for the prevention of CL-ABI that represent a collaborative effort by a multidisciplinary coalition of professional organizations that provide evidence based recommendations to prevent catheter related infections [5]. The interventions emphasize five distinct practices, including: education and training of healthcare providers who place and care for catheters, utilizing maximum sterile barrier precautions during catheter placement, skin preparation using 2% chlorhexidine, avoiding routine replacement of central lines as a strategy to reduce infection, and using antiseptic or antibiotic coated lines in the event that infection rates remain high despite adherence to the above measures [5].

Several studies have demonstrated impressive reductions in CL-ABI from the application of these strategies, ranging from 18 to 100% reductions and realizing significant reductions in mortality and cost [2]. The simple introduction of maximum sterile barrier precautions to insert central lines has been observed to dramatically reduce infection rates for over a decade [6]. However, the CDC's guidelines, despite their seeming simplicity, have been found to be frequently insufficiently applied, whether by ignorance or omission (2) In the past 12 months there have been a total 24 documented central venous catheter (CVC) infections at SLRHC. At RH the total number of central line days since June 2005 was3,567 with a cumulative rate of infection of 2.8 per 1000 central line days and at SLH a total of 8,524 central line days with an infection rate of 4.3 per 1000 central line days. These infection rate figures are above the benchmark experience. The cost of CVC infections to hospitals in the United States is estimated to be $45,000 per infection (7). For SLRHC the cost incurred over the past 12 months is estimated to be $1,080,000.

Training and education of healthcare personnel and the utilization of maximum sterile precautions are two important areas. Residents still most frequently learn central line placement techniques by the "see one, do one, teach one" method, which by its very definition allows for a multitude of techniques in practice. While this teaching theoretically includes the utilization of maximal sterile precautions for central line placement, the focus of teaching, and of residents' anxieties, is most often focused on the proper placement of the line, not the sterile technique used to place it. Residents in non-surgical fields may not be comfortable with maximum sterile technique in bedside procedures, and surgical residents may be somewhat blasé about the need for such detail.

Medical simulators allow residents to practice skills in a realistic and interactive environment that minimizes risk to patients. Studies have found simulation to be an effective means for teaching skills as diverse as ACLS and airway management to laparoscopic surgical skills (8, 9, 10). Additionally, the use of audio-visual equipment in a medical simulator to record a resident's performance gives valuable firsthand feedback that is otherwise not available, as it allows residents to visualize their own missteps (11). This is hypothesized to be of particular value in the proper acquisition of physical skills such as maximum sterile precautions.

We plan to examine the utility of a medical simulation environment that replicates an ICU setting to first assess medical residents' ability to utilize and maintain maximum sterile precautions in the placement of central venous lines using a standardized scoring tool and subsequently, assess the impact of videotape training vs. individual simulated debriefing on performance of correct MBP.

We hypothesize that medical residents, who have baseline training in the placement of central venous lines, will show improvement following simulation and viewing of the training videotape, and that greatest improvement will be seen in the residents who go through a debriefing simulated method. We hypothesize that PGY 2 and 3 medical residents undergoing simulation-based training in maximal barrier precaution technique during central venous catheter (CVC) placement will have good recall after 3 months

ELIGIBILITY:
Inclusion Criteria:

* Medical residents who completed one year training in internal medicine program who are certified by their program to place and supervise medical interns in placement of CVC

Exclusion Criteria:

* Refusal to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: MEDICAL RESIDENTS
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
-Primary outcome: Medical residents' performance in maximal barrier precaution (MBP) technique during central venous catheter (CVC) placement | 2 weeks

SECONDARY OUTCOMES:
Secondary outcome: Medical residents' confidence level in maximal barrier precaution (MBP) technique during CVC placement | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Khouli, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St. Luke's Roosevelt Hospital, New York, New York, United States

REFERENCES:
- [Derived] Khouli H, Jahnes K, Shapiro J, Rose K, Mathew J, Gohil A, Han Q, Sotelo A, Jones J, Aqeel A, Eden E, Fried E. Performance of medical residents in sterile techniques during central vein catheterization: randomized trial of efficacy of simulation-based training. Chest. 2011 Jan;139(1):80-7. doi: 10.1378/chest.10-0979. Epub 2010 Aug 12. PMID 20705795